CLINICAL TRIAL: NCT05679804
Title: Turkish Validity and Reliability Study of The Bipolar Recovery Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Zehra GÜNAY YAĞCI, Assistant Professor, Bilecik Seyh Edebali Universitesi
Other Study IDs: BilecikSeyhEU
Record Dates: First submitted 2022-12-24; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Bipolar Disorder, Recovery
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: validity and realibility of scale — Turkish validity and realibility of Bipolar Recovery Questionnare

SUMMARY:
In addition to objective criteria (no episode period for 6 months) for defining and monitoring recovery, evaluation of subjective criteria is also very important. Various Turkish scales related to recovery in progressive diseases have been developed or validity-reliability studies have been conducted. However, as far as we know, there is no scale that evaluates subjective improvement for a disorder such as bipolar disorder that progresses in episodes and has a heterogeneous appearance of loss of functionality. In this study, we aimed to conduct a validity and reliability study of the recovery questionnaire for BDD.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 ages
* Be diagnosed with bipolar affective disorder
* Be at least primary school graduate

Exclusion Criteria:

* having a physical disability (blindness, etc.) that might prevent filling in the scales,
* having an additional neurological disease that prevented filling out the scale items.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bipolar Affective Disorder
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-04-13 (Estimated); Study Completion 2023-05-13 (Estimated)

PRIMARY OUTCOMES:
validity and reability of scale | 5 months
  turkish validity and reability of Bipolar Recovery Questionnare

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Seyh Edebali University Faculty of Medicine, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No